CLINICAL TRIAL: NCT02664428
Title: Measuring the Impact of Dietary Supplementation With New Baking Product PreBIOil on Gut Microbiota and Cholesterol Metabolism
Brief Title: Measuring the Impact of Dietary Supplementation With a New Baking Product on Gut Microbiota and Cholesterol Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Edmund Mach (Other)
Collaborators: Casa di Cura Eremo di Arco (TN) Italy (Unknown); OlioCRU Consorzio srl Arco (TN) Italy (Unknown)
Responsible Party: Principal Investigator, Kieran Tuohy, Dr, Fondazione Edmund Mach
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PreBIOil 2
Record Dates: First submitted 2016-01-16; First posted 2016-01-27 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREBIOIL TEST (Active Comparator): Product tests prepared with olives flour, buckwheat flour, pea flour, chestnut flour, oil chemical leavening agents, salt, sucrose. Baked
  Interventions: Dietary Supplement: PreBIOil
- CONTROL (Placebo Comparator): Product control prepared with wheat flour, oil, chemical leavening agents, salt, sucrose. Baked
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: PreBIOil — A daily dose of about 90 gram will be given for 8 weeks
  Arms: PREBIOIL TEST
Dietary Supplement: Control — A daily dose of about 90 gram will be given for 8 weeks
  Arms: CONTROL

SUMMARY:
Study hypothesis: Diet integrated with food prepared with olive, buckwheat, peas and chestnut flour as in PreBIOil product combination can modify the gut microbiota and the cholesterol metabolism.

Primary objectives of the study are to assess whether the test product to be able to change:

1. fecal microbiota profile;
2. Plasma cholesterol LDL, total, total LDL and HDL ratio;
3. plasma triglycerides;
4. Apolipoprotein ApoA-I, ApoB, and Lp.

Secondary objectives of the study are:

1. anthropometric indices;
2. secondary metabolites of polyphenols in human biofluids;
3. mass spectrometry plasma and urine metabolite profile;
4. blood glucose and fasting insulin levels; 5,6) C-reactive protein (PRC or hsPRC);

7) urinary isoprostane F2; 8) oxidized LDL in plasma.

Study Design: placebo-controlled, randomized, double-blind parallel trial.

Inclusion criteria: Aged 30-65 years; BMI 20-29,9 kg/m^2. Total Cholesterol 180-240 mg/dl

Exclusion criteria: Fasting blood glucose >150 mg/dl; triglycerides >500 mg/dl; uncontrolled hypertension (blood pressure [BP] >160/100 mm Hg under antihypertensive therapy); any long term medical therapy; food intolerances; alcohol intake >5 drinks per day or use of narcotic substances; use of dietary supplements, pro or pre- biotics; special diet; pregnancy, tobacco smoking.

Methodology: Determination of eligibility: for each volunteer aged between 30 and 65 years, will undergo to clinical and biochemistry evaluation. Clinical visit, clinical tests, and blood drawing will be performed after an overnight fasting at visit T-1 at the Casa di Cura Eremo di Arco (TN). In this T-1 visit the eligibility will be established and the participants will be randomized to receive supplementation with either PreBIOil biscuit (90g/day) or Control for 8 weeks in a double-blind manner. Clinical tests, blood drawing, and stool and urine collection will be performed during visits at the beginning and end of each treatment period (T0 and T1). A 4 day-food diary record will be collected before visits T0, at the beginning of T0 and before T1.

Efficacy Assessments Arterial BP; BMI; ratio of waist to hip circumference; food questionnaires; blood sample analysis (total cholesterol, triglycerides, HDL and LDL cholesterol, oxidized LDL, serum glucose and insulin, C-RP, Apolipoproteins, Isoprostane; urinary and plasma metabolite profiling; fecal microbiota analysis.

Safety assessments. Adverse events registration.

Statistical analyses. The differences between the two group will be evaluated with univariate and multivariate statistical methods. The medium before and after the intervention will be compared with the General Linear Model (ANOVA) for repeated measures or for paired data. Simple and multiple linear regressions will be performed to determine the relationships between independent variables; also we will run the t-test to evaluate differences in compliance detected in the types of supplementation. The results are expressed as mean +/- SEM and the differences will be considered significant when P <0.05.

Duration: Subjects will make three visits (visit T-1, beginning visit T0, and end of treatment period visit T1, week 8 from T0). The treatment duration is 8 weeks; a daily portion of about 90 g of biscuit is introduced.

DETAILED DESCRIPTION:
The first results of in vitro testing of the project PreBIOil have delineated the capacity of a flour of olives to modulate the microbial population of the human intestine in a manner comparable to that of inulin recognized as polysaccharide with a capacity prebiotic. Based on these results, and to others in the literature, the bakery product PreBIOil has been formulated. The product contains, flour of olives, buckwheat, pea, and chestnut.

The overall objective of the study is to assess whether the introduction in the diet of a bakery product prepared with olive flour, mixed with buckwheat, pea and chestnuts flour can change the profile of the intestinal microbiota and the plasma cholesterol, in particular LDL. The study is set up as dietary supplementation, double-blind, randomized, parallel with the control group, in which the following product will be compared:

i) a new bakery product designed study PreBIOil (test); ii) a bakery product control isoenergetic (control).

Description of the Food supplemented in the Trial The test product is new baked product formulated with a mixture of flour from olives, buckwheat, pea and chestnut and has the appearance of a salty biscuit.

Participants will be required to consume daily about 90 grams of test or control product. The exact quantities of each product batch will be determined following the assessment of the nutritional characteristics of the finished product in order to provide the same calorie intake with the two products.

Digestibility, fermentability and modulation of the microbiota Buckwheat is considered a non-cereal that in addition to containing fiber, minerals and vitamins, such as B2 and B6, also represents a source of antioxidant compounds due to the content of flavonoids.

The pea flour contains important components for human diet (starch, protein and other nutrients). The health benefits associated with consumption of peas primarily derived from the concentration and properties of starch, protein, fiber, vitamins, minerals and phytochemicals. The fiber contained in the integument and in the cell walls of the cotyledon contributes to gastrointestinal function. The starch content in pea flour is characterized by lower glycemic index. The proteins from pea may produce peptides with antioxidant activity. The vitamin and mineral content of peas can play an important role in the prevention of deficiency diseases, in particular those relating to the deficiencies of selenium and folate. Peas contain a variety of phytochemicals. These include polyphenols that may have antioxidant and anticancer, saponins which are present hypo colesterolemica and anticancer activities, and oligosaccharides of galactose that can exert prebiotic benefits in the large intestine.

The nutritional components of chestnut flour consist of carbohydrates, protein and fat in the composition such as to provide an energy value about 350-400 kcal / 100 g. Chestnuts have been voted to have a positive effect on the metabolism of gut bacteria and are a source of long-chain fatty acids C18: 1 and C18: 2 and vitamins (vitamin E). The possible presence of polyphenols is limited to the outer skins, generally separated from the fruit during the production of the flour. The flour coming from olive paste is not described in the scientific literature for specific nutritional properties for the human diet. However olives are an integral part of the Mediterranean diet in which they are consumed as table olives and olive oil. The olive fruit contains 50% water, 22% fat, about 19% of carbohydrates and about 2% of protein; the polyphenol content varies in the range 1-3%. The olives are consumed or as olive oil or table olives. The olives are characterized by strong bitterness, caused mostly dall'oleuropein. The oleuropein can reach 140 mg / g dry weight in unripe olives and decreases and as the fruit ripens Table olives are treated to mitigate the bitter taste through processes such as maceration soda and fermentation in brine. However in the process of sweetening the bitterness over lost some important compounds present in olives such as polyphenols and fiber. There is no evidence on the ability of extra virgin olive oil polyphenols reducing the risk of cardiovascular disease, but a large part of the possible effects of the components of the olive alone or in synergy with the polyphenols are still unexplored. In addition a large part of the water-soluble fraction contained in the olives, between which the fibers and polyphenols with proven beneficial activities on human health, is not removed in the process of oil production. There is evidence that some phenolic fractions as secoiridoids are poorly absorbed by the intestinal mucosa and are then available for the colonic microflora. Essentially the oil in its entirety would have the greatest potential as a food can modulate beneficially the composition and activity of microorganisms symbiotic human gut, as observed experimentally for other types of fruit.

By means of simulation in vitro of colonic fermentation it has been observed that the olive paste, even after baking at 180°C for 30 ', is capable of modulating the human intestinal microbiota with a prebiotic effect or inducing a significant increase of bifidobacteria. Such simulation in vitro was carried out by incubation for 24 h in a batch fermentation system with control of pH and temperature, following inoculation with feces obtained from five healthy individuals. The analysis of total polyphenols (main antioxidants present in the test product) present in the flour of olives, in the mixture of the flour and in the test product did detect a loss of total polyphenols, as a result of baking equal to 40%.

Clinical Results Clinical results have shown that daily consumption of 100 g of buckwheat in the form of flour has determined the increase in the HDL/cholesterol ratio and improved glucose tolerance and more recently it was observed that the consumption of biscuits made of buckwheat has reduced the serum level of a marker of inflammation, myeloperoxidase (MPO) in addition to a reduction of total cholesterol with better pulmonary vital capacity. A recent meta-analysis of several intervention studies on the human diet with supplementation of legumes, including peas, showed their ability to decrease serum levels of LDL cholesterol.

Intervention studies on diet with olive oils, by-products of processing of olives and olive-based products have been conducted with healthy volunteers and subjects with various degrees of cardiovascular risk. Of these studies have been indicated the daily doses of total polyphenols introduced (from a few mg / day to 30 mg / day, up to 100 mg / day) depending on the type of olive oil and also enrichment with extracts. These interventions had in many cases a duration of about a month, and most of the studies measured the effects of antioxidant and anti-inflammatory changes in the circulatory system, along with the values of plasma lipids, and other parameters related to oxidative stress. In particular in the study "EUROLIVE", on a large sample of healthy individuals, it was observed that the phenols of olive oil were able to protect blood lipids from oxidation, increase the concentration of HDL cholesterol and the relationship between reduced and oxidized glutathione, however no changes dell'F2-isoprostane.

In 2011 the European Food Safety Authority (EFSA) has approved the claim that the olive oil polyphenols, especially hydroxytyrosol, protect LDL from oxidation, at a dose greater than or equal to 5 mg/kg/day. Other studies have also shown that olive oil polyphenols are related to the reduction of CRP, reduced atherogenic gene expression in blood cells, and decreased blood pressure. Although there are evidences on the ability of olive oil polyphenols to reduce the risk of cardiovascular diseases, a large part of the possible effects of the components of the olive alone or in synergy are still unexplored. Moreover, a large part of fibers and polyphenols contained in the olive is not extracted in the process of oil extraction and eliminated as a byproduct.

Rationale of the Study The buckwheat flour adds fiber and flavonoids, the pea flour contains carbohydrates with low glycemic index, protein and is also a source of antioxidants, chestnut flour brings prebiotic substances and vitamins. Flour olive is the fruit of the olive is with its water-soluble components (eg. Fibers and polyphenols) and in the soluble fraction of polyunsaturated and monounsaturated fatty acids, tocopherols and carotenoids that only partially pass extra virgin olive. These components are designed mostly as components of extra virgin olive oil and scientifically have given evidence to contribute to the improvement of lipid metabolism and plasma lipids framework, to heart health and protect against oxidative stress.

Based on available clinical and experimental studies, it has been suggested that consumption of a baked product made from a mixture of flour from olive paste, buckwheat, peas and chestnuts can have positive effects on lipid plasma biomarkers and intestinal microbiota (for example, an increase of bifidobacteria) in adult participants with plasma content of cholesterol in medium to high levels even if not yet pathological.

Statement of compliance statement This study will be carried out in compliance with the Protocol and in accordance with Good Clinical Practice (GCP), as described in ICH GCP for 1996, the US Code of Federal Regulations (CFR) and the Declaration of Helsinki. With the signing of this protocol, the researcher agrees to comply with these requirements.

Objectives of the study

The overall objective of the study is to assess whether the introduction in the diet of a new bakery product containing a mixture of flour from olive paste, buckwheat, peas, chestnuts is able to change:

Primary objectives:

1. The profile of fecal microbiota;
2. Plasma levels of total cholesterol, LDL, ratio / total LDL and HDL;
3. The plasma levels of triglycerides;
4. Apolipoprotein ApoA-I, ApoB, and Lp (a).

Secondary objectives:

1.The anthropometric indices 2 The secondary metabolites of polyphenols in human biofluids 3.The profiles of metabolites in plasma and urine assessed by analysis of mass spectrometry (MS); 4. The blood glucose and fasting insulin levels; 5. C-reactive protein (PRC); 6. High-sensitivity C-reactive protein (hsPRC); 7. urinary isoprostane F2; 8. oxidized LDL in plasma.

Presentation experimental design Participants volunteers will be identified and recruited at an outpatient part of the Casa di Cura Eremo di Arco (TN). Participants will be informed about the purposes and methods of the study and will be pre-selected based on criteria for inclusion / exclusion. The participant, will sign the informed consent and will enter the studio after the visit to T-1, performed at outpatient part of Casa di Cura Eremo di Arco (TN) where it will be performed a clinical and biochemical health status. To allow proper monitoring of eating habits, the eligible participant, after the first visit will fill a food diary.

If subjects will be eligible for the study based on all the criteria for inclusion and exclusion, will be randomized to receive either placebo or the active integration at visit T0.

The clinical examination, and the collection of blood and urine will be carried out after fasting for about 10 hours at the beginning of the start-up period (visit T-1). Clinical tests, blood samples, collection of feces and urine will be performed during visits T0, T1. Additional food diary (4 consecutive days) will be filled at visits T0 and ahead of T1. Adverse events, taking medications and supplements will be recorded by the participants in a special diary.

Participants included in the study will also be asked to fill in a sensory evaluation of each food offered in blind, the first taste and at the end of 8 weeks of supplementation for each product

Study Procedure Recruitment of participants Participants will be identified and recruited at an outpatient part of Casa di cura Eremo di Arco (TN) Participants will be informed about the purposes and methods of the study and will be pre-selected based on criteria for inclusion/exclusion. If eligible, the participant will sign the informed consent and will enter the studio with a visit to T-1, which will be performed during a clinical and biochemical state of health. The subjects that will be eligible for the study based on all the criteria for inclusion/exclusion, will be included in the study and randomized to receive the first food supplementation (test or control) to visit T0 (two weeks later by the run-in).

Supplementation

After eligibility is assessed, the participants will be randomized to receive the integration with the bakery product with the test or control product:

The single daily doses will be packaged in packs encoded by a qualified group. Supplementation will last eight weeks, double-blind, parallel. with one of the two products (attributed to randomization).

Follow up The project will consist of a period of eight weeks of supplementation, clinical examinations and the collection of blood and urine will be made after an overnight fast (excluding water consumption) of about 10 hours to visit T-1 . Clinical tests, blood collection, the collection of feces and urine tests will be carried out visits to T0, T1: T0 is the day of the first integration, T1 will be eight weeks after the start of treatment. The food diary will be compiled to visit T-1 and distributed before visits T0 and T1 for data collection visits T0 and T1.

Clinical evaluation Electrocardiogram. An ECG will be performed at screening (T-1). The ECG tracings will be reviewed and interpreted by the outpatient part of the nursing home Hermitage of Arco.

Blood pressure will be measured according to the guidelines for hypertension ISH / WHO 2004 Anthropometric indices Weight and height will be measured on a standard scale. The measures will be carried out on subjects without shoes, coats or warm clothes. Body-mass index, BMI, is calculated as kg /m2.

The waist circumference (umbilical) will be measured in a manner determined by the National Institutes of Health, National Heart, Lung, and Blood Institute.The ratio of the circumference of the waist and hip ratio (WHR) is calculated.

Questionnaires All information will be collected and recorded in validated questionnaires, including personal identification, medical history and information on the risk factors for cardiovascular disease, medication use, physical activity and eating habits. Also a four-day food diary will be written by each participant.

Participants included in the study will also be asked to fill in a sensory evaluation of each food offered in the first blind tasting and at the end of 8 weeks of supplementation.

Sampling of blood and urine collection The blood (≤ 30 ml) will be drawn from a peripheral vein, after 10 hours of fasting. 24 h urine will be collected, the volume measured and sample will be stored at -80 ° C.

Collection of fecal samples Fecal samples will be processed within 12 hours of sample collection. Aliquots of each fecal sample will be frozen directly at -80 ° C for analysis of metabolomic profile.

Laboratory tests by the laboratory analysis of the Casa di Cura Eremo di Arco Blood samples will be centrifuged according to the requirements of the tests to be performed immediately after blood collection. Plasma or serum will be separated, in part immediately tested and the remaining fraction stored at -80 ° C.

Total cholesterol, HDL cholesterol, triglycerides and glucose will be evaluated with enzymatic method. LDL cholesterol will be measured analytically with enzymatic method.

Insulin levels will be assessed by elettrochemioluminescenza. The blood count and platelet count will be assessed by method impedentiometric. The C-reactive protein (CRP) will be measured by turbidimetric assay. The high-sensitivity C-reactive protein (hsPCR) will be measured by turbidimetric assay.

Apolipoprotein AI (ApoA-I), ApoB, and Lp (a) were determined by immunoturbidimetry.

The test for the verification of the absence of glucosuria will be made by measuring the concentration of glucose in the urine.

Laboratory tests by the Fondazione Edmund Mach [EMF] Urinary and plasma metabolomic profile. The F2-isoprostanes will be measured in the urine as a measure of oxidative stress, by means of specific EIA kit, after purification by chromatography solid phase (columns SepPack).

The analysis of LDL oxidized in the plasma will be conducted with the aid of ELISA kit.

The samples of urine and blood (plasma and serum) will be subjected both to analysis of targeted metabolomics (UPLC-MS / MS for non-volatile compounds and GC-MS / MS for volatile compounds) that analyzes of non-targeted metabolomics (ULPC-Q -TOF-MS and Nano -FTMS-Q-TOF nonvolatile and GC-TOF for the volatile compounds). For profiles of targeted plasma metabolites, it will be used the MS-based Biocrates AbsoluteIDQ ® Kit P180, generating precise quantitative data on 180 human metabolites linked to the risk of diabetes. In addition, specific targeted analysis will be applied to the lipid profile of serum bile acids, short-chain fatty acids (short chain fatty acids, SCFAs) and quantification of metabolites of the polyphenols of microbial origin in biofluids (including feces) with UPLC / QQQ-MS / MS.

Analysis of fecal microbiota. Changes in the faecal microbiota of specific bacterial populations will be evaluated using the method of in situ hybridization with fluorescent probes (FISH).

Also changes in the faecal microbiota will be evaluated using a metagenomics approach using pyrosequencing 454. In short, after the collection of stool samples (n = 128, 2 stool samples at different times T0, T1 from 64 subjects before and after consumption of each food test and placebo) will extract the bacterial genomic DNA using the kit SPIN FastDNA (MPbio) specific for feces. Using primers specific for the bacterial 16S rRNA gene (hypervariable region V1-V3) it will be performed by PCR amplification and then subjecting the amplified V1-V3 at 454 pyrosequencing.

Will use the GS FLX Titanium Chemistry with adapters Multiplex Identifier (MID) to get sequences of length 600 bp that will be analyzed by comparing the database of 16S rRNA phylogenetic, publicly available, via the pipeline QIIME that allows assignment to the genus level of human intestinal microbiota. It will be produced a total of about 20,000 sequences for each fecal sample. As quality control and analysis of microbial ecology, it will be used a multivariate statistical in order to correlate the changes in the composition of the fecal microbiota following the consumption of food testing or placebo.

Randomization blinded Participants will be assigned randomly but equally distributed by sex and age to one of two treatments: bakery product test or control product even using specific software. The clinical researchers, investigators and laboratory personnel will be blinded to the randomization.

Treatment The supplementation will be introduced in the daily diet through the consumption of a bakery product (test) for a daily consumption of 90 grams of product containing flour of olives, from buckwheat, from peas, chestnuts. The food will provide an analogue control calorie intake. The products under study (test or control) will be supplied in packs that will be labeled in the local language with the code number of the study. the manufacturer's name, the number of patients, the number of study visit. The products will be distributed to the participants from the visit T0.

Duration of study and planning After eligibility will be assessed, participants will be randomized in two groups (product test or control) that will follow 8 weeks of dietary supplementation.

The overall duration of the study, including the start-up period (run-in) and the treatment will be 10 weeks.

The recruitment will start later and within three months of approval by the Ethics Committee.

The run-in will begin within two weeks of the first visit (T-1). Subjects will be recruited over a period of 10 months and the study will be completed within 12 months from the time of the first recruitment.

Criteria for study discontinuation In accordance with the Declaration of Helsinki, ICH standards of good clinical practice, and the "Food and Drug Administration (FDA) Regulations" of the United States, a person has the right to withdraw from the study at any time and for any reason, without prejudice for future medical care from the physician or the institution. Investigators also have the right to withdraw the study subjects (see below). In the event that a person (or a person legally authorized representative) decides to retire, every effort will be made to complete and report the observations as well as possible. A final comprehensive assessment should be made at the time of the withdrawal of the subject where the reason for the withdrawal must be registered and in any case should an attempt be made to perform a follow-up evaluation.

The Subjects can be removed from the study for the following reasons:

Breach of the Protocol as from the experimenter Not meaningful compliance by the subject The refusal of the subject to continue treatment or comments Unacceptable toxicity Decision of the researcher that the closure is in the best medical interest of the subject Unclear event of illness or complications Use of concomitant medications that are incompatible with the study. Pregnancy Abuse of alcohol or drugs Those who discontinue or is withdrawn from the study will not be replaced.

Procedure for Terminating

If an individual stop before the completion of the study, the reason and the cutoff date will be recorded. The date of the last dose of food in the study should be recorded. In the event of early termination, the following procedures must be performed:

Clinical tests (systolic and diastolic, heart rate, weight and height to calculate BMI and waist and hip circumference).

Taking blood and feces and urine collection. A food frequency questionnaire (weekly). In the event that the individual can not return for follow-up visit, the investigators will have groped to contact the person by phone to track any adverse events.

If a person withdraws consent to receive food in the studio, you will be encouraged to remain in the study without receiving treatment for the collection of safety data.

The procedures of reliability of the product under study The products (test or control) will be provided in packages labeled in the local language with the code number of the study, the number of site code, the manufacturer's name, the number of participants, the number of visits of the study, the number of lot, instructions for storage and expiration dates. The products will be distributed to the participants from the visit T0.

Codes randomization The codes of randomization by sex and age, for each participant will be stored in a sealed envelope by qualified group of Sensory Quality (QS of the Department of Nutrition and Food Quality of the Research and Innovation Centre of the Edmund Mach Foundation).

Data Source Control All data collected during the study will be obtained from primary sources, and will be recorded in written documents and electronic medical records as the subject. The results of clinical, laboratory results and ECG will be recorded in the electronic medical record file of the subject. No data will be inserted directly in the "case report form" (CRF), without being transferred from the primary source, such as paper records or electronic.

Concomitant Drug Therapy Any medication taken from the subject within one month before the start of the study and / or administered during the study will be considered as concomitant therapy. Such treatment must be documented on the appropriate page of the CRF and the medical records of the subjects. Any changes to the concomitant therapy during the study must be clearly recorded and the reason for the change should be documented.

A letter will be sent to the doctor of each participant, specifying what are the treatments concomitant incompatible with the study. The use of the following drugs will not be allowed during the study: blood thinners, antihypertensives, lipid-lowering drugs, beta-blockers, systemic corticosteroids, neuroleptics, antibiotics, laxatives, vitamin supplements, antioxidants and minerals, dietary fiber, prebiotics (eg inulin, oligofructose) and probiotics. Therefore if the subject requires drug therapies incompatible with the study, the subject is notified by the treating physician to terminate the study and inform the head of the study and following the procedures for the early termination.

Compliance Rating To assess compliance to supplementation, they will be measured urinary phenols in subjects that will be supplemented with food tests at T0, T1. In addition, all the unused or empty packaging at the end of each week will be returned to the experimenters.

Methods Security There were no security problems during previous studies related to the consumption of products made from olives, buckwheat, pea flour, chestnut flour.

The study will be monitored by medical and paramedical staff of the Casa di Cura Eremo of Arco. Adverse events will still be recorded throughout the study. Abnormal laboratory values that induce clinical signs or symptoms or require therapeutic intervention will be promptly notified to the subject, if the subject has explicitly expressed that wish to receive such communication in the form of informed consent. The subject will be free to withdraw from the study in advance if in need of therapeutic intervention is not compatible with the study, or if you experience adverse events that cause a change in the criteria for inclusion of this subject in the study. The subject will still be free to withdraw from the study at any time, in case the study is due to discomfort following the procedure for early termination.

Statistical analysis The basic features are listed by type of supplementation: continuous variables are expressed as mean +/- standard deviation or medians with interquartile ranges and as a percentage for categorical variables. Data with an asymmetric distribution will follow a log processing prior to analysis. The differences between the two supplements will be evaluated with univariate and multivariate statistical methods. The medium before and after the intervention will be compared with the General Linear Model (ANOVA) for repeated measures or for paired data. You will perform simple and multiple linear regressions to determine the relationships between independent variables; also we will run the test to evaluate differences in compliance detected in the types of supplementation. The results are expressed as mean +/- SEM and the differences will be considered significant when P <0.05. Data with an asymmetric distribution will follow a log processing prior to analysis.

The main analysis will be based on a comparison of the differences in mean levels after consumption of test product and after consumption of control. The differences between the mean values at the end of each supplementation (T1) in relation to the relative mean baseline value (T0) will also be measured.

The differences in time between treatment arms will be evaluated by analysis of variance for repeated measures.The level of significance will be considered <0.05 in two tails.

The sample size for each supplementation has been determined to 32 to detect a decrease of LDL cholesterol in the plasma equal to about 15.44 mg/dl with a standard deviation of 14.28 mg/dl using the equation Snedecor and Cochran with α equal to 0.05 and 1-β equal to 0.9 (Dell et al., 2002). According to this formula the minimum number of subjects to enroll is equal to 28. Taking into account possible dropouts, 32 people for supplementation with the test product and 32 people for supplementation with control product for a total of 64 volunteer subjects in this study.

The assessment is made on the basis of the abundance of the decrease of LDL cholesterol in plasma, on the basis of the measures (mean and standard deviation) of LDL cholesterol reported in a parallel study published in the European Journal of Nutrition. The parameter LDL cholesterol, in addition to being an effect on human health recognized is more restrictive and requires observation times longer than the extent of the modification of the intestinal microflora.

Direct access to source data / documents Regulatory authorities may wish to carry out checks on clinical research to evaluate compliance with the principles of GCP. Regulatory authorities may also wish to conduct an inspection (during the trial or after its completion). If an inspection required by a regulatory authority and / or the Ethics Committee for Clinical Trials c/o APSS Trento, the researcher must agree to provide access, regulatory authorities, the documentation related to the study.

Data Management and Records The source of the data and documentation is defined as the first place where the data is recorded. Any original documents and should not be kept and made available at the same location. The researcher must keep the original documents for each person participating in the study.

The data collected on the CRF during the trial will be documented in an anonymous way, and those will be identified by numbers or symbols. If in exceptional circumstances it is necessary, for reasons of safety or regulation, identifying the person, OlioCRU Ltd and the researcher are required to keep such information confidential.

All data entered in the CRF shall be legible and recorded in black ink. Should you require a correction it should be made by deleting the entry with a single line and entering the correct information next to the item itself. The correction must be initialed and dated by the investigator, or a qualified person designated.

ELIGIBILITY:
Inclusion Criteria:

* male and female;
* age between 30 and 65 years;
* with BMI (body mass index, BMI) of between 20 and 29.9 kg/m2,
* total plasma cholesterol in the range 180-240 mg/dl.

Exclusion Criteria:

Subjects will be excluded from participation in the study if they meet one of the following exclusion criteria:

* fasting glucose> 140 mg/dl;
* triglycerides> 500 mg/dl;
* uncontrolled hypertension (BP >160/100 mm Hg under antihypertensive therapy); cardiovascular disease (myocardial infarction, percutaneous transluminal coronary angioplasty or coronary artery bypass grafting, unstable angina pectoris, stoke, peripheral arterial disease);
* hypo or hyperthyroidism;
* acute inflammatory diseases;
* serious gastrointestinal disease;
* hypo- or hyperthyroidism;
* acute inflammatory diseases;
* severe gastrointestinal diseases;
* heart, liver, renal or pulmonary failure or other life threatening disease with prognosis <5 years;
* chronic use of systemic corticosteroids, anti-coagulants, anti-inflammatory, or lipid lowering and anti-diabetics drugs;
* treatment within the previous 6 weeks with any medication that is known to affect lipoprotein levels or fecal microbiota (specifically, antibiotics);
* food intolerances;
* alcohol intake >5 drinks per day or use of narcotic substances;
* use of antioxidant vitamin or mineral supplements;
* special diet;
* pregnancy;
* smoking.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Faecal microbiota analysis | 8 weeks
  Faecal microbiota analysis by FISH and 454 Roche pyrosequencing

SECONDARY OUTCOMES:
Cholesterol Metabolism | 8 weeks
  Analysis of total, LDL, HDL cholesterol in plasma
Triglycerides | 8 weeks
  Analysis of plasma levels of triglycerides
Apolipoproteins | 8 weeks
  Apolipoprotein ApoA-I, ApoB, and Lp (a) analysis in plasma

OTHER OUTCOMES:
The anthropometric indices | 8 weeks
  Analysis of the variation of the anthropometric indices
The secondary metabolites of polyphenols in human biofluids | 8 weeks
  Analysis of the polyphenols secondary metabolites in human biofluids
Urine metabolites profile | 8 weeks
  Measuring profiles of metabolites in plasma and urine assessed by analysis of mass spectrometry (MS)
Plasma metabolites profiles | 8 weeks
  Meauring the profiles of metabolites in plasma assessed by analysis of mass spectrometry (MS)
Fasting insulin levels | 8 weeks
  Analysis asting insulin levels
Blood glucose | 8 weeks
  Analysis of the blood glucose
C-reactive protein (PRC) | 8 weeks
  Analysis of C-reactive protein (PRC)
Urinary isoprostane F2 | 8 weeks
  Analysis of urinary isoprostane F2
Oxidized LDL in plasma | 8 weeks
  Analysi of oxidized LDL in plasma
Faecal Bile Acids | 8 weeks
  MS analysis of fecal bile acid concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Viola, PhD, Study Director — Fondazione Edmund Mach
Locations (2):
- Italy (2):
  - Casa di Cura Eremo, Arco, Trento
  - Centro Ricerca Innovazione Fondazione Edmund Mach, San Michele all'Adige, Trento